CLINICAL TRIAL: NCT03548441
Title: Comparative Effectiveness and Prognostic Factors for Outcome of Surgical and Non-surgical Management of Lumbar Spinal Stenosis in an Elderly Population: Protocol for an Observational Study
Brief Title: Comparative Effectiveness and Prognostic Factors of Surgical and Non-surgical Management of Lumbar Spinal Stenosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Spine Centre of Southern Denmark (Other)
Collaborators: University of Southern Denmark (Other); Parker Research Institute (Other); Odense University Hospital (Other); University College South Denmark (Other); University of Aarhus (Other); Defactum, Central Denmark Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 17/30636
Record Dates: First submitted 2018-04-30; First posted 2018-06-07 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery: Exposed
  Interventions: Procedure: Surgery
- Non-surgical management: Non-exposed
  Interventions: Other: Non-surgical management

INTERVENTIONS:
Procedure: Surgery — Patients receiving surgical treatment undergo various types of posterior decompressive surgery with or without spinal fusion. The method used for decompressive surgery or fusions is determined solely by the surgeon.
  Groups: Surgery
Other: Non-surgical management — Patients managing lumbar spinal stenosis non-surgically are either referred to rehabilitation primary health care center or referred back to their general practitioner for treatment. Treatment may include physiotherapy, chiropractic treatment, lifestyle changes and/or pain management. Post-surgically patients may also be referred to rehabilitation at a primary health care center.
  Groups: Non-surgical management

SUMMARY:
Introduction: Lumbar spinal stenosis is a common cause of low back and leg pain in elderly impacting physical activity and quality of life. Initial treatments are non-surgical options. If unsuccessful, surgery is advocated. The literature is not clear as to the outcome of surgery when compared to non-surgical treatment, and the optimal time for surgery is not explicit.

Materials and analysis: This observational study is designed to investigate the course of treatment, compare effectiveness of surgical and non-surgical treatment in patients with lumbar spinal stenosis, and identify prognostic factors for outcome in the context of current clinical practice. Prospectively registered data on treatment, outcome and patient characteristics are collected from nationwide registers on health and social issues, a clinical registry of people with chronic back pain and hospital medical records. Primary outcome is change in physical function measured by the Zurich Claudication Questionnaire. Secondary outcomes are changes in symptom severity, pain-related function, health-related quality of life, and general self-efficacy. All outcomes are measured at baseline, 6 months and 12 months follow up. Comparisons on these variables will be made between those who undergo surgery for lumbar spinal stenosis and those not receiving surgery at 12 months follow up according to different analysis populations. Prognostic factors include treatment allocation, back and leg pain intensity, comorbidity, duration of symptoms, pre-treatment function, self-rated health, income, general self-efficacy and magnetic resonance imaging graded compression of central stenosis.

Ethics and dissemination: The study has been evaluated by The Regional Committees on Health Research for Southern Denmark (S-20172000-200) and notified to the Danish Data Protection Agency (17/30636). All participants provide consent. Findings will be disseminated in peer-reviewed publications and presented at national and international conferences following the guidance from the STROBE and PROGRESS statement. Potential sources of bias will be addressed using ROBINS-I.

ELIGIBILITY:
Inclusion Criteria:

1. >60 years.
2. ICD-10 diagnosis of degenerative lumbar spinal stenosis registered in the nationwide patient registry between January 1st - December 31st 2017.
3. Included in the SpineData registry.
4. Give consent to use patient-reported data for research purposes

Exclusion Criteria:

-

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >60 years, diagnosed with lumbar spinal stenosis and having first clinical contact at the Spine Center of Southern Denmark, Hospital Lillebaelt, Middelfart from January 1st - December 31st 2017 eligible for this study, will be identified in the National Patient Register. Follow-up time from the date of first clinical contact (baseline) is 6 and 12 months.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Physical function | Between baseline and 12 months follow up
  Change in physical function score in the Zurich Claudication Questionnaire (ZCQ) collected through a clinical registry of people with chronic back pain (SpineData).
  The ZCQ is a condition-specific self-reported measure of symptom severity, physical function and satisfaction with treatment in patients with lumbar spinal stenosis.
  The questionnaire is composed of three domains (subscales) with a Likert-type scale.
  The physical function subscale includes 6 items addressing walking distance and walking ability. All but one item have Likert response scales with 4 categories.
  The physical function subscale score is calculated from the unweighted mean of all answered items.
  The possible range of the score is 1 to 4.
  Lower scores indicate less disability.

SECONDARY OUTCOMES:
Symptom severity | Between baseline and 12 months follow up
  Change in symptom severity score in the Zurich Claudication Questionnaire (ZCQ) collected through a clinical registry of people with chronic back pain (SpineData).
  The ZCQ is a condition-specific self-reported measure of symptom severity, physical function and satisfaction with treatment in patients with lumbar spinal stenosis.
  The questionnaire is composed of three domains (subscales) with a Likert-type scale.
  The symptom severity subscale includes 7 items addressing pain, numbness, weakness and balance disturbances. All but one item have Likert response scales with 5 categories.
  The possible range of the score is 1 to 5.
  Lower scores express less symptom severity.
Pain related physical function | Between baseline and 12 months follow up
  Change in Oswestry Disability Index collected through a clinical registry of people with chronic back pain (SpineData).
  The Oswestry Disability Index (ODI) is a region-specific questionnaire for assessing self-reported levels of disability for patients with spinal disorders.
  The questionnaire contains 10 pain related sections (items) with 6 response options (statements). Each section of six response options is scored from 0 (no pain) to 5 (most severe pain).
  For each section of six statements the total score is 5; if the first statement is marked, the score equals 0; if the last (6th) statement is marked, the score equals 5. If more than one box is marked in each section, the highest score is used.
  The section scores are summarised to a total score, ranging from 0-100. Scores are expressed as a percentage of total points.
  Lower scores indicate less disability.
Health related quality of life | Between baseline and 12 months follow up
  Change in health related quality of life measured by EQ-5D-3L collected through a clinical registry of people with chronic back pain (SpineData).
  The EQ-5D-3L is a generic self-reported instrument for measuring health-related quality of life consisting of a descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression), each with 3 response options.
  These are converted into a single summary index by applying preference weights obtained from the general population with a total score ranging from -0.6 to 1, where 1 corresponds to perfect health and 0 to death.
  Higher scores indicate better health related quality of life,
  The EQ VAS is a vertical, visual analogue scale scoring patients self-rated health ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
  Higher scores indicate better self-perceived health.
General self-efficacy | Between baseline and 12 months follow up
  Change in general self-efficacy score obtained by the General Self Efficacy Scale collected through a clinical registry of people with chronic back pain (SpineData).
  The General Self efficacy scale is a self-reported unidimensional measure of general sense of perceived self-efficacy designed for the general adult population and used in patients with chronic pain.
  The questionnaire comprises of 10 items (statements) with 4 response options. Responses are scored on a 4-point Likert-scale from 1 (not true at all) to 4 (exactly true).
  Responses of all 10 items are summarised to yield the final composite score with a range from 10 - 40 points.
  Higher scores express greater perceived self-efficacy.

OTHER OUTCOMES:
Diagnosis | At baseline
  ICD-10 diagnosis codes collected from nationwide registers
Age | At baseline
  Potential prognostic factor / confounder collected from nationwide registers
Sex | At baseline
  Potential prognostic factor / confounder collected from nationwide registers
Height | At baseline
  Potential prognostic factor / confounder collected through a clinical registry of people with chronic back pain (SpineData)
Weight | At baseline
  Potential prognostic factor / confounder collected through a clinical registry of people with chronic back pain (SpineData)
Cohabitation status | At baseline
  Potential prognostic factor / confounder collected from nationwide registers
Income | At baseline
  Potential prognostic factor / confounder collected from nationwide registers
Socio-economic classification | At baseline
  Potential prognostic factor / confounder collected from nationwide registers
Work status | At baseline
  Potential prognostic factor / confounder collected from nationwide registers
Highest level of education completed | At baseline
  Potential prognostic factor / confounder collected from nationwide registers
Number of consultations in primary health care centers | From baseline to 12 months follow up
  Potential prognostic factor / confounder collected from nationwide registers
Number of hospital admissions | From baseline to 12 months follow up
  Potential prognostic factor / confounder collected from nationwide registers
Use of prescriptive analgesic medicine | From baseline to 12 months follow up
  Potential prognostic factor / confounder collected from nationwide registers
Hospital department | From baseline to 12 months follow up
  Potential prognostic factor / confounder collected from nationwide registers
Duration of symptoms | At baseline
  Potential prognostic factor / confounder collected through a clinical registry of people with chronic back pain (SpineData)
Low back pain intensity | From baseline to 12 months follow up
  Change in Numerical Pain Rating Scale (NPRS) as Potential prognostic factor / confounder collected through a clinical registry of people with chronic back pain (SpineData).
  The Numeric Pain Rating Scale (NPRS) is an 11-point, unidimensional measure of pain intensity in which patients rate their pain ranging from 0 (no pain) to 10 (worst pain imaginable).
  Lower scores indicate less pain.
Leg pain intensity | From baseline to 12 months follow up
  Change in Numerical Pain Rating Scale (NPRS) as potential prognostic factor / confounder collected through a clinical registry of people with chronic back pain (SpineData).
  The Numeric Pain Rating Scale (NPRS) is an 11-point, unidimensional measure of pain intensity in which patients rate their pain ranging from 0 (no pain) to 10 (worst pain imaginable).
  Lower scores indicate less pain.
Comorbidity | From baseline to 12 months follow up
  Charlson comorbidity index as potential prognostic factor / confounder collected from nationwide registers.
  The Charlson Comorbidity Index is a method of categorising comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes found in administrative data, such as a national patient registry.
  Each comorbidity category has an associated weight (from 1 to 6), based on the relative risk of 1-year mortality. The sum of all the weights results in a single comorbidity score for a patient.
  An index score of 0 indicates that no comorbidities were found.
  A higher index score indicates a higher risk of death within 1 year.
Degree of central stenosis | At baseline
  Potential prognostic factor / confounder collected from Magnetic Resonance Imaging (MRI) descriptions in hospital medical records.
  MRI graded compression is estimated using a classification ranging from mild to moderate or severe stenosis.
  Mild stenosis is defined as narrowing of one-third of the normal area or less, moderate stenosis as narrowing of between one- and two-thirds, and severe stenosis as narrowing of more than two-thirds of the area.

CONTACTS AND LOCATIONS:
Overall Officials: Helle A Brøgger, MSc, Principal Investigator — 1) Spine Centre of Southern Denmark, 2) University of Southern Denmark, 3) The Parker Research Institute, 4) University College South Denmark; Robin Christensen, PhD, Study Director — 1) The Parker Research Institute 2) Odense University Hospital; Thomas Maribo, PhD, Study Director — 1) Aarhus University 2) DEFACTUM; Berit Schiøttz-Christensen, PhD, Study Chair — 1) Spine Centre of Southern Denmark, 2) University of Southern Denmark
Locations (1):
- Spine Centre of Souther Denmark, Middelfart, Fyn, Denmark

REFERENCES:
- [Derived] Brogger HA, Maribo T, Christensen R, Schiottz-Christensen B. Comparative effectiveness and prognostic factors for outcome of surgical and non-surgical management of lumbar spinal stenosis in an elderly population: protocol for an observational study. BMJ Open. 2018 Dec 19;8(12):e024949. doi: 10.1136/bmjopen-2018-024949. PMID 30573489